CLINICAL TRIAL: NCT02402530
Title: A Randomized, Double-blind Trial Investigating the Efficacy and Safety of Intravenous Neridronic Acid in Subjects With Complex Regional Pain Syndrome Type I (CRPS-I)
Brief Title: Efficacy and Safety of Intravenous Neridronic Acid in CRPS-I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF7013-01; U1111-1151-2181 (Other: World Health Organization); 2014-001915-37 (EudraCT Number)
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Complex Regional Pain Syndrome, Type I
Keywords: Neridronic Acid; Neridronate; CRPS; RSD
MeSH Terms: conditions — Reflex Sympathetic Dystrophy | interventions — 6-amino-1-hydroxyhexane-1,1-diphosphonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo administered as intravenous infusion on Day 1, Day 4, Day 7 and Day 10
  Interventions: Drug: Placebo
- 125 mg Neridronic acid (Experimental): Neridronic acid 62.5 mg administered as intravenous infusion on Day 1 and Day 4; matching placebo administered as intravenous infusion on Day 7 and Day 10
  Interventions: Drug: Placebo; Drug: Neridronic acid 62.5 mg
- 250 mg Neridronic acid (Experimental): Neridronic acid 62.5 mg administered as intravenous infusion on Day 1, Day 4, Day 7 and Day 10
  Interventions: Drug: Neridronic acid 62.5 mg

INTERVENTIONS:
Drug: Placebo — Matching placebo administered as intravenous infusion.
  Arms: 125 mg Neridronic acid; Placebo
Drug: Neridronic acid 62.5 mg — Neridronic acid administered as intravenous infusion.
  Arms: 125 mg Neridronic acid; 250 mg Neridronic acid

SUMMARY:
This clinical trial is being conducted to demonstrate the efficacy of neridronic acid in the treatment of pain associated with complex regional pain syndrome type I (CRPS-I).

The trial is divided into 3 periods: a 60-day enrollment period, a 12-week trial period, and an extended follow-up period with visits at Month 6, Month 9, and Month 12. The extended follow-up period will be terminated for all participants after the last participant enrolled completes their Month 6 visit (Visit 9). The double-blind will be maintained throughout the 12-week trial period and extended follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed.
* Male or female participant between 18 years and 80 years of age.
* A diagnosis of complex regional pain syndrome type I according to the clinical diagnostic criteria using the International Association for the Study of Pain clinical diagnostic criteria (Budapest criteria).
* Baseline Pain Intensity Score of 4 or greater using an 11-point Numerical Rating Scale referring to the CRPS-affected limb.
* In stable treatment and follow-up therapy for CRPS type I for at least 1 month.
* Participant has undergone a recent regular dental examination.
* Women of child-bearing potential must have a negative urine ß-HCG pregnancy test at enrollment.
* Women of child-bearing potential must practice protocol defined acceptable methods of birth control during the trial.
* Participants must be able to communicate meaningfully, be able to differentiate with regard to location and intensity of the pain, and be able to answer the questions in the questionnaires used in this trial.
* Compliance with the use of electronic diary assessed prior to allocation to treatment.

Exclusion Criteria:

* A diagnosis of complex regional pain syndrome type II.
* Documented history or diagnosis of peripheral neuropathy, including diabetic peripheral neuropathy or other metabolic or toxic neuropathy, or any other chronic pain condition that would significantly affect a participant's ability to report CRPS-related pain.
* Body weight less than 40 kg.
* Evidence of renal impairment or a history of chronic kidney disease.
* Serum calcium or magnesium outside of the central laboratory's reference range; history of hypocalcemia; any metabolic disorder anticipated to increase risk for hypocalcemia.
* Vitamin D deficiency. Participants with vitamin D deficiency prior to enrollment may be enrolled with appropriate supplementation during the enrollment period.
* Corrected QT interval greater than 470 milliseconds; treatment with medications within the last 30 days prior to allocation to IMP that have potential to prolong the QT interval or anticipated need for such medications during the course of the trial.
* Any prior use of a bisphosphonate for treatment of CRPS, any prior administration of intravenous bisphosphonate, administration of oral bisphosphonate within the previous year, anticipated requirement for treatment with oral or intravenous bisphosphonate for another condition such as osteoporosis during the trial, or administration of denosumab (Prolia) or other bone turnover suppressing drugs within the past 6 months.
* History of any allergic or hypersensitivity reaction to neridronic acid or other bisphosphonate, or to vitamin D or calcium supplements.
* Recent tooth extraction, unhealed or infected extraction site, or significant dental/periodontal disease that may pre-dispose to need for tooth extraction or other invasive dental procedures during the trial.
* Evidence of denture-related gum trauma or improperly fitting dentures causing injury.
* Prior radiation therapy of the head or neck (within 1 year of enrollment).
* Recent treatment with high doses of systemic steroids or anticipated need for concomitant high-dose steroid treatment during the trial.
* History of malignancy within 2 years before enrollment with the exception of basal cell carcinoma.
* Daily intake of long- and short-acting or controlled-release opioid analgesics of more than 200 mg morphine equivalents, regimens combining high-dose opioids and benzodiazepines, or any other treatment regimen considered unstable, unsafe, or have potential to affect the interpretation of the trial.
* Use of nerve blocks, ketamine infusions, intravenous immunoglobulin, acupuncture, electromagnetic field treatment, or initiation/implementation of radiofrequency ablation or other sympathectomy procedures, or peripheral nerve stimulation within 6 weeks prior to allocation to investigational medicinal product.
* Evidence of current alcohol or drug abuse, or history of alcohol or drug abuse within 2 years of enrollment, based on participant history and physical examination and according to the investigator's judgment.
* Any other severe medical condition, including severe depression, or any other severe mood disorder, that in the opinion of the investigator may affect efficacy or safety assessments or may compromise the participant's safety during trial participation.
* Participant is engaged in litigation related to their disability from CRPS in which monetary gain or loss (or other compensation) may affect their objective participation in the trial.
* Women who are pregnant or breastfeeding.
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2-fold upper limit of normal (ULN), or evidence or history of liver disease.
* Participation in an investigational drug trial within 3 months prior to enrollment, or prior participation in this trial with receipt of any infusion of IMP, even a partial infusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in the Pain Intensity Score to Week 12. | Baseline; Week 12
  The Pain Intensity Score is the mean value of current pain intensity ratings, obtained twice-daily for 1 week, using an 11-point numerical rating scale where 0 = "no pain" and 10 = "pain as bad as you can imagine". All pain intensity ratings for the primary endpoint will be in reference to the CRPS-affected limb.

SECONDARY OUTCOMES:
Response to treatment: Proportion of Participants With at Least 30 Percent Reduction in the Pain Intensity Score | Baseline; Week 12
  Participants with at least a 30 percent decrease in the Pain Intensity Score will be considered to have responded to treatment. The Pain Intensity Score is determined as for the primary endpoint.
Response to treatment: Proportion of Participants With at Least 50 Percent Reduction in the Pain Intensity Score | Baseline; Week 12
  Participants with at least a 50 percent decrease in the Pain Intensity Score will be considered to have responded to treatment. The Pain Intensity Score is determined as for the primary endpoint.
Change in the Brief Pain Inventory (BPI) Interference Score | Baseline; Week 12
  The BPI Interference Score is the mean value of 7 self-reported items in question 9 of the BPI Short Form Questionnaire. Participants will rate their interference of pain with general activity, walking, work, sleep and other activities in the past 24 hours, with possible ratings from 0 (does not interfere) to 10 (completely interferes). The BPI interference Score ranges from 0 to 10, with higher values indicating greater pain interference of daily activities.
Patient Global Impression of Change (PGIC) | Baseline; Week 12
  The PGIC is a self-reported measure of perceived change in overall condition since the start of the study. Participants will select one of seven responses ranging from very much improved to very much worse. A response of very much improved or much improved is generally regarded as a clinically important outcome.
Change in the EuroQol-5 Dimension 5 Level (EQ-5D-5L) Index Score | Baseline; Week 12
  The EQ-5D-5L Index Score describes the participant's overall health status and is derived from self-reported scores in 5 health dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Participants will rate each dimension at one of 5 levels, with level 1 indicating the best health state (no problems) and level 5 indicating worst health state (e.g., unable to walk about). The EQ-5D-5L Index Score ranges from 0 to 1, with 0 representing death and 1.0 representing perfect health.
Change in the EuroQol Visual Analog Scale (EQ VAS) | Baseline; Week 12
  The EQ VAS is a self-reported measure of the participant's overall health "today". Participants will place a mark on a 20 cm vertical scale numbered from 0 to 100, with 0 labeled as "the worst health you can imagine" and 100 labeled as "the best health you can imagine". The EQ VAS ranges from 0 to 100, with higher scores representing better overall health.

OTHER OUTCOMES:
Change in the Worst Pain Intensity | Baseline; Week 12
  This will be determined as for the primary endpoint, using worst pain intensity ratings. Participants will rate their worst pain intensity during the previous 12 hours twice each day using an 11-point numerical rating scale where 0 = "no pain" and 10 = "pain as bad as you can imagine". Worst pain intensity ratings are in reference to the CRPS-affected limb.
Change in the Average Pain Intensity | Baseline; Week 12
  This will be determined as for the primary endpoint, using average pain intensity ratings. Participants will rate their average pain intensity during the previous 12 hours twice each day using an 11-point numerical rating scale where 0 = "no pain" and 10 = "pain as bad as you can imagine". Average pain intensity ratings are in reference to the CRPS-affected limb.
Change from Baseline in the Pain Intensity Scores at Each Week | Baseline to Week 12
  Pain Intensity Scores will be determined as for the primary endpoint using current pain intensity ratings obtained twice-daily. Mean values will be assessed during each of the first 12 weeks of the study.
Response to Treatment: Proportion of Participants with 0 to 100% Decrease in the Pain Intensity Score | Baseline; Week 12
  Pain Intensity Scores will be determined as for the primary endpoint using current pain intensity ratings obtained twice-daily. Participants will be considered to have responded to treatment using increments of 10% decrease in the Pain Intensity Score, starting from 0% (no decrease in the Pain Intensity Score), 10%, 20%, etc., to 100% (Pain Intensity Score at Week 12 = 0).
Response to Treatment: Proportion of Participants With at Least a 2 Point Decrease in the Pain Intensity Score | Baseline; Week 12
  Pain Intensity Scores will be determined as for the primary endpoint using current pain intensity ratings obtained twice-daily. Participants will be considered to have responded to treatment if they have at least a 2 point decrease in the Pain Intensity Score.
Change in the Pain Anxiety Symptom Scale (PASS) Total Score | Baseline; Week 12
  The PASS Total Score is the sum of 20 self-reported items in the PASS Questionnaire. Participants will rate each item in terms of its frequency, ranging from 0 (never) to 5 (always). The PASS Total Score ranges from 0 to 100, with higher scores indicating greater levels of pain-related anxiety.
Change in the Center for Epidemiological Studies Depression (CES-D) Scale Total Score | Baseline; Week 12
  The CES-D Total Score is the sum of 20 self-reported items comprising symptoms associated with depression. Participants will rate each item in terms of its frequency from "rarely or none of the time (less than 1 day)" to "most or all of the time (5 to 7 days)" during the last week. The CES-D Total Score ranges from 0 to 60, with a score over 21 indicating the possibility of major depression.
Change in Pain Disability Index (PDI) | Baseline; Week 6; Week 12
  The PDI is the sum of self-reported ratings of disability in 7 categories of activities, including family/home responsibilities, recreation, social activity, self-care, etc. Participants will rate the level of disability that they typically experience due to pain in each of the 7 categories. Ratings are made using a numeric rating scale, with 0 indicating "no disability" and 10 indicating "worst disability". The PDI ranges from 0 to 70, with higher values indicating greater disability due to pain.
Change in the Medical Outcomes Study (MOS) Sleep Scale: Sleep Problems Index | Baseline; Week 6; Week 12
  The MOS Sleep Scale Sleep Problems Index is derived from participant's responses to questions related to sleep adequacy, sleep disturbance, daytime somnolence, and other aspects of sleep. Participants will respond to 12 questions in the MOS Sleep Scale Questionnaire. Responses are scored, summed and converted to a 0 to 100 scale, with higher scores indicating worse sleep problems.
Change in Pain Medication Score | Baseline; Week 6; Week 12; Month 6; Month 9; Month 12
  The Pain Medication Score will be derived using the Medication Quantification Scale (MQS III) and is based entirely on information available from the participant's prior and concomitant medications. The MQS III algorithm derives a single numerical value representing the amount of pain medications taken by each participant, taking into account the medication class and dosage.
Change in the Current Pain Intensity in the Extended Follow-up Period | Baseline; Month 6; Month 9; Month 12
  Participants will rate their current CRPS-related pain intensity at each visit in the extended follow-up period using an 11-point numerical rating scale where 0 = "no pain" and 10 = "pain as bad as you can imagine".
Change in the Average Pain Intensity in the Extended Follow-up Period | Baseline; Month 6; Month 9; Month 12
  Participants will rate their average CRPS-related pain intensity, recalled over the last 24 hours, at each visit in the extended follow-up period using an 11-point numerical rating scale where 0 = "no pain" and 10 = "pain as bad as you can imagine".
Change in the Worst Pain Intensity in the Extended Follow-up Period | Baseline; Month 6; Month 9; Month 12
  Participants will rate their worst CRPS-related pain intensity, recalled over the last 24 hours, at each visit in the extended follow-up period using an 11-point numerical rating scale where 0 = "no pain" and 10 = "pain as bad as you can imagine".
Change in the BPI Interference Score in the Extended Follow-up Period | Baseline; Month 6; Month 9; Month 12
  The BPI Interference Score is the mean value of 7 self-reported items in question 9 of the BPI Short Form Questionnaire. Participants will rate their interference of pain with general activity, walking, work, sleep and other activities in the past 24 hours, with possible ratings from 0 (does not interfere) to 10 (completely interferes). The BPI interference Score ranges from 0 to 10, with higher values indicating greater pain interference of daily activities.
PGIC in the Extended Follow-up Period | Baseline; Month 6; Month 9; Month 12
  The PGIC is a self-reported measure of perceived change in overall condition since the start of the study. Participants will select one of seven responses ranging from very much improved to very much worse. A response of very much improved or much improved is generally regarded as a clinically important outcome.
Change in the EQ-5D-5L Index Score in the Extended Follow-up Period | Baseline; Month 6; Month 9; Month 12
  The EQ-5D-5L Index Score describes the participant's overall health status and is derived from self-reported scores in 5 health dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Participants will rate each dimension at one of 5 levels, with level 1 indicating the best health state (no problems) and level 5 indicating worst health state (e.g., unable to walk about). The EQ-5D-5L Index Score ranges from 0 to 1, with 0 representing death and 1.0 representing perfect health.
Change in the EQ VAS in the Extended Follow-up Period | Baseline; Month 6; Month 9; Month 12
  The EQ VAS is a self-reported measure of the participant's overall health "today". Participants will place a mark on a 20 cm vertical scale numbered from 0 to 100, with 0 labeled as "the worst health you can imagine" and 100 labeled as "the best health you can imagine". The EQ VAS ranges from 0 to 100, with higher scores representing better overall health.
Change in the Complex Regional Pain Syndrome (CRPS) Severity Score | Baseline; Week 6; Week 12; Month 6; Month 9; Month 12
  The CRPS Severity Score is the sum of the number of CRPS-related symptoms, reported by the participant over the past 48 hours, and signs, observed by the clinician during a brief examination. Participants are queried for 8 CRPS-related symptoms and assessed for 8 CRPS-related signs, for a score between 0 and 16, with higher scores indicating greater CRPS severity.
Presence or Absence of Complex Regional Pain Syndrome (CRPS) | Month 6; Month 9; Month 12
  The presence or absence of CRPS will be determined based on CRPS-related signs, assessed by the clinician in a brief examination. Participant reported symptoms for CRPS from the Enrollment Visit will be included with signs applying the CRPS diagnostic criteria ("Budapest clinical criteria"). Participants who meet criteria for CRPS using the diagnostic criteria will be considered as "CRPS present", and those who do not meet the criteria will be considered as "CRPS absent".
Change from Baseline in Bone Turnover Markers | Baseline to Month 12
  Serum levels of bone formation markers (procollagen type I amino-terminal propeptide and bone alkaline phosphatase) and a bone resorption marker (C-terminal telopeptide of type I collagen) will be determined from blood samples taken during the trial. This information will be used for an exploratory evaluation of bone turnover in response to neridronic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (59):
- United States (49):
  - Site US119 - G & L Research, Foley, Alabama
  - Site US117 - Valley Pain Consultants, Scottsdale, Arizona
  - Site US116 - Arizona Pain Specialists, Scottsdale, Arizona
  - Site US124 - Quality of Life Medical and Research Centers LLC, Tucson, Arizona
  - Site US154 - Woodland International Research Group, Little Rock, Arkansas
  - Site US110 - Orange County Research Institute, Anaheim, California
  - Site US172 - Core Healthcare Group, Cerritos, California
  - Site US108 - Catalina Research Institute, Chino, California
  - Site US175 - Inland Pain Medicine, Colton, California
  - Site US152 - UC San Diego Healthcare Systems, Center for Pain Medicine, La Jolla, California
  - Site US102 - Samaritan Center for Medical Research, Los Gatos, California
  - Site US126 - Northern California Research, Sacramento, California
  - Site US106 - Mountain View Clinical Research, Denver, Colorado
  - Site US153 - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Site US162 - South Lake Pain Institute, Clermont, Florida
  - Site US143 - Florida Pain Institute, Merritt Island, Florida
  - Site US111 - Sunrise Research Institute, Miami, Florida
  - Site US122 - Precision Research Organization, LLC, Miami Lakes, Florida
  - Site US104 - Discovery Clinical Trials, Orlando, Florida
  - Site US133 - Gold Coast Research LLC, Plantation, Florida
  - Site US171 - Florida Medical Pain Management, St. Petersburg, Florida
  - Site US121 - Clinical Research of West Florida, Tampa, Florida
  - Site US165 - Palm Beach Research, West Palm Beach, Florida
  - Site US131 - Better Health Clinical Research, Inc, Newnan, Georgia
  - Site US103 - Great Lakes Clinical Trials, Chicago, Illinois
  - Site US129 - International Clinical Research Institute, Overland Park, Kansas
  - Site US169 - Massachusetts General Hospital, Boston, Massachusetts
  - Site US127 - Advance Clinical Research, Inc, St Louis, Missouri
  - Site US105 - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Site US101 - Princeton Medical Institute, Princeton, New Jersey
  - Site US151 - Premier Pain Centers, Shrewsbury, New Jersey
  - Site US156 - University Clinical Research Center, Somerset, New Jersey
  - Site US166 - Albany Medical College, Albany, New York
  - Site US145 - University of Rochester, Rochester, New York
  - Site US137 - Montefiore Medical Center, The Bronx, New York
  - Site US135 - The Center for Clinical Research, Winston-Salem, North Carolina
  - Site US157 - North Star Medical Research, Middleburg Heights, Ohio
  - Site US149 - Founders Research Corporation, Philadelphia, Pennsylvania
  - Site US114 - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Site US112 - Clinical Trials of South Carolina, Charleston, South Carolina
  - Site US107 - Austin Center for Clinical Research, Austin, Texas
  - Site US134 - Lovelace Scientific Resources, Inc, Austin, Texas
  - Site US113 - Pioneer Research Solutions, Inc, Houston, Texas
  - Site US118 - Omega International Pain Clinic, Salt Lake City, Utah
  - Site US164 - Advanced Clinical Research, West Jordan, Utah
  - Site US144 - Bellevue Surgery Center, Bellevue, Washington
  - Site US173 - Bellevue Surgery Center, Bellevue, Washington
  - Site US123 - Northwest Clinical Research Center, Bellevue, Washington
  - Site US161 - Swedish Pain and Headache Center, Seattle, Washington
- Germany (5):
  - Site DE107 - Studienzentrum A. Schwittay, Böhlen
  - Site DE104 - Schmerzzentrum Dr. med. C. Wachter & T. Tusker, Fellbach
  - Site DE101 - Klinische Forschung Hannover Mitte GmbH, Hanover
  - Site DE103 - Algesiologikum Studienzentrum und Algesiologikum MVZ, Munich
  - Site DE102 - Universitätsklinikum Würzburg Neurologische Klinik, Würzburg
- United Kingdom (5):
  - Site GB104 - The Royal Victoria Infirmary, Cambridge
  - Site GB108 - Darlington Memorial Hospital, Centre for Research and clinical Intervention, Darlington
  - Site GB109 - Royal Devon Exeter Hospital, Exeter
  - Site GB101 - Guys and St. Thomas NHS Foundation Trust - St Thomas Hospital, London
  - Site GB111 - Chelsea and Westminster Hospital - NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details); according to the EFPIA Data Sharing Principles.
URL: http://www.grunenthal.com/r-d-vision-mission/pipeline/data-sharing-clinical-trials